CLINICAL TRIAL: NCT01429662
Title: Phase 3 Study of Modified Relaxation (MR) Technique for Treating Hypertension in Postmenopausal Women
Brief Title: Modified Relaxation (MR) Technique for Treating Hypertension in Postmenopausal Women
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chiang Mai University (Other)
Responsible Party: Principal Investigator, Suprawita Saensak, PhD candidate (Clinical Epidemiology), Chiang Mai University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MRLE-HTN
Record Dates: First submitted 2011-09-03; First posted 2011-09-07 (Estimated); Last update posted 2012-05-30 (Estimated); Status verified 2012-05

CONDITIONS: Postmenopausal Syndrome; Hypertension
Keywords: postmenopause; hypertension; relaxation; SBP 140-159 mmHg; DBP 90-99 mmHg; stage 1 or mild hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lifestyle Education (LE) (Sham Comparator): Lifestyle Education (LE) Participants in this group will receive conventional care and lifestyle education on dietary choice and exercise.
  Interventions: Behavioral: Lifestyle Education (LE)
- Modified Relaxation (MR) (Experimental): Modified Relaxation (MR) This technique intend to train participants in a group of 8-10 in only 1 session that lasts 60 minutes. After completing the training, participants will be given a hand-out on MR. They will be asked to practice MR at home once a day for 15-20 minutes during their leisure times, for at least 5 days a week during the whole 16 weeks of the study period.
  Interventions: Behavioral: Modified Relaxation (MR)

INTERVENTIONS:
Behavioral: Modified Relaxation (MR) — Modified Relaxation (MR) This technique intend to train participants in a group of 8-10 in only 1 session that lasts 60 minutes. After completing the training, participants will be given a hand-out on MR. They will be asked to practice MR at home once a day for 15-20 minutes during their leisure times, for at least 5 days a week during the whole 16 weeks of the study period.
  Other Names: Behavioral Relaxation
  Arms: Modified Relaxation (MR)
Behavioral: Lifestyle Education (LE) — Participants in this group will receive conventional care and lifestyle education on dietary choice and exercise.
  Other Names: Lifestyle Modification
  Arms: Lifestyle Education (LE)

SUMMARY:
The purpose of this study is to demonstrate better effectiveness of modified relaxation (MR) technique over no MR for treating hypertension in Thai postmenopausal women.

DETAILED DESCRIPTION:
Medical treatment of hypertension (HTN) in postmenopausal women is not very effective, as it requires co-operation and long-term commitment from the patients and their families. The medication itself may cause bothersome side effects and it can pose economic burden to the patients and the society. In contrast, lifestyle modifications, particularly relaxation technique, are less costly and relatively free of any side effects. Once the patients master the techniques, they can practice by themselves at home and at any time that is convenient to them. There is evidence from at least one RCT that the techniques are effective in reducing the systolic blood pressure (SBP) and diastolic blood pressure (DBP), even after a short practice of only two months.

In this study, the investigators propose a randomized control trial to examine the effectiveness of modified relaxation (MR) technique to control HTN in Thai postmenopausal women against a control group who practice no MR. Such a study in Thai population has not been done before. In addition, the investigators will extend the period of observation up to 16 weeks, to assess longer-term patients' compliance, and the effects of MR on BP.

ELIGIBILITY:
Inclusion Criteria:

* Stage 1 essential hypertension, defined as a systolic blood pressure of 140-159 and/or DBP of 90-99 mmHg on two occasions at least 30 minutes apart.
* Women who are able to attend follow visits as advised.

Exclusion Criteria:

* Women with systolic blood pressure (SBP) >160 mmHg or diastolic blood pressure (DBP) >100 mmHg.
* Women who have other known causes of hypertension, such as renal diseases
* Women who are using sedatives or tranquilizer,or antidepressant, or antihypertensive medication during the past 2 months prior to the study.
* Have language or geographical barrier.
* Do not give their informed consent.
* Women who need to be prescribed HRT.

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 429 (Actual)
Dates: Start 2011-08; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Changes in SBP. | 16 weeks
  Measure the systolic blood pressure (SBP) after intervention at 1, 2 ,3 , and 4 months.

SECONDARY OUTCOMES:
Changes in DBP. | 16 weeks
  Measure the diastolic blood pressure (DBP) after intervention at 1, 2 ,3 , and 4 months.
Continuation rate of MR practice. | 16 weeks
  Measure the continuation rate of MR practice after 4 months of follow-up period.
Drop-out rates. | 16 weeks
  Measure the drop-out rate after intervention at 1, 2, 3, and 4 months of follow-up period.
Numbers of subjects who require anti-hypertensive medication. | 16 weeks
  Measure the numbers of subjects who require anti-hypertensive medication after intervention 4 months of follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Suprawita Saensak, PhDcandidate, Principal Investigator — PhD in Clinical Epidemiology Program, Faculty of Medicine, Chiang Mai University (Thailand)
Locations (1):
- Mahasarakham Hospital, Maha Sarakham, Northeast, Thailand

REFERENCES:
- [Derived] Saensak S, Vutyavanich T, Somboonporn W, Srisurapanont M. Modified relaxation technique for treating hypertension in Thai postmenopausal women. J Multidiscip Healthc. 2013 Oct 3;6:373-8. doi: 10.2147/JMDH.S51580. eCollection 2013. PMID 24124377
- See also: NIH is the nation's medical research agency-supporting scientific studies that turn discovery into health. — http://www.nih.gov
- See also: PubMed comprises more than 21 million citations for biomedical literature from MEDLINE, life science journals, and online books. — http://www.ncbi.nlm.nih.gov/pubmed
- See also: The Journal of North American Menopause Society is a peer-reviewed scientific journal owned by NAMS and published by Lippincott Williams & Wilkins (LWW). — http://www.menopause.org
- See also: The Journal of Behavioral Medicine is a broadly conceived interdisciplinary publication devoted to furthering understanding of physical health and illness through the knowledge and techniques of behavioral science. — http://www.springer.com/medicine/journal/10865